CLINICAL TRIAL: NCT05078112
Title: Clinical Testing of a Novel Device to Promote Sleep Continuity in Infants
Brief Title: Sleep Device Testing to Promote Sleep in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103800
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sleep Device intervention (Experimental): Infants will utilize the sleep device during sleep for 20 days
  Interventions: Device: Sleep sensor technology

INTERVENTIONS:
Device: Sleep sensor technology — Infants will sleep on a novel device with built-in sensor technology that tracks sleep patterns and provides output to soothe them to sleep. The device will give this output for first 10 nights, then wean the output the child receives over 10 nights.

SUMMARY:
Infants often have sleep challenges. Most of these challenges in otherwise healthy children and due to behavioral insomnia. The goal for infants is to become independent sleepers by learning the process of self-soothing. This study hopes to determine if technology based on sensors is able to help teach self-soothing to infants.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 2-12 months.
2. Meets clinical criteria for behavioral insomnia of childhood, sleep association subtype, as defined by the International Classification of Sleep Disorders Manual.

Exclusion Criteria:

1. Diagnosed comorbid health problem that may disrupt sleep.
2. History of birth prior to 37 weeks gestational age.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sujay Kansagra, MD, Principal Investigator — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Duke Pediatric outpatient clinics from October 2021 to June 2022.
Groups:
- Sleep Device Intervention: Infants will utilize the sleep device during sleep for 20 days.
  Infants will sleep on a novel device with built-in sensor technology that tracks sleep patterns and provides output to soothe them to sleep. The device will give this output for first 10 nights, then wean the output the child receives over 10 nights.
Period: Overall Study
Arm/Group | Sleep Device Intervention
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sleep Device Intervention
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Nighttime Awakenings Per Night as Measured by Parent Sleep Diary
Description: Parents reported number of nighttime awakenings on the 5 days immediately prior to intervention (at baseline) and 5 days immediately following the intervention. The intervention takes place during the 20 days in between the measurement of baseline measures and post-intervention measures. The number of nighttime awakenings is averaged over the 5 days prior to intervention and compared to the average over 5 days after intervention.
Time Frame: Baseline to 5 days post-intervention
Measure: Mean (Standard Deviation); unit: awakenings per night
Arm/Group | Sleep Device Intervention
Number analyzed (Participants) | 19
awakenings per night | -0.88 (0.89)
Statistical Analysis 1: Comparison: Sleep Device Intervention; Test type: Other; p = 0.000393, t-test, 2 sided

2. Secondary Outcome: Change in BISQ-SF (Brief Infant Sleep Questionnaire - Short Form) Score
Description: The BISQ-SF is a research tool that measures infant sleep metrics, parental perceptions of the child's sleep, and parental behaviors. The total score is scaled from 0 to 100, with higher scores denoting better sleep quality, more positive perception of infant sleep, and parent behaviors that promote healthy and independent sleep.
Time Frame: Baseline to post-intervention (approximately 20 days)
Population: Caregivers were not considered enrolled, but did contribute to this assessment. Each caregiver that had pre and post-intervention BISQ-SF scores available contributed to this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Device Intervention
Number analyzed (Participants) | 34
score on a scale | 13.4 (10.6)

3. Secondary Outcome: Change in Caregiver Epworth Sleepiness Scale (ESS)
Description: Caregivers evaluate their own sleepiness via the ESS. The ESS has a total score range of 0 to 24, where a higher score indicates greater sleepiness.
Time Frame: Baseline to post-intervention (approximately 20 days)
Population: Caregivers were not considered enrolled but did contribute to this assessment. Each caregiver that had pre and post-intervention ESS scores available contributed to this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Device Intervention
Number analyzed (Participants) | 34
score on a scale | -0.94 (2.95)

4. Secondary Outcome: Change in Patient Health Questionnaire-2 (PHQ-2) Score
Description: A PHQ-2 score ranges from 0 to 6, where a higher score indicates a greater frequency of depressed mood and anhedonia.
Time Frame: Baseline to post-intervention (approximately 20 days)
Population: Caregivers were not considered enrolled but did contribute to this assessment. Each caregiver that had pre and post-intervention PHQ-2 scores available contributed to this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sleep Device Intervention
Number analyzed (Participants) | 34
score on a scale | -0.47 (1.16)

ADVERSE EVENTS:
Time Frame: Approximately 20 days
Arm/Group | Sleep Device Intervention
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT05078112/Prot_SAP_000.pdf